CLINICAL TRIAL: NCT02533843
Title: Outcome of Different Ablation Strategies In Persistent and Long-Standing Persistent Atrial Fibrillation
Acronym: OASIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCAI_OASIS
Record Dates: First submitted 2014-12-05; First posted 2015-08-27 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I (Active Comparator): ablation at sources guided by FIRMap (using RhythmView™ Workstation from TOPERA) Intervention: AF ablation
  Interventions: Procedure: radiofrequency catheter ablation
- Arm II (Active Comparator): ablation at sources guided by FIRMap (using RhythmView™ Workstation from TOPERA) + conventional pulmonary vein antrum isolation (PVAI) Intervention: AF ablation
  Interventions: Procedure: radiofrequency catheter ablation
- Arm III (Active Comparator): Extended PVAI plus ablation of non-PV triggers and complex fractionated atrial electrograms (CFAE) Intervention: AF ablation
  Interventions: Procedure: radiofrequency catheter ablation

INTERVENTIONS:
Procedure: radiofrequency catheter ablation — Radiofrequency catheter ablation of atrial fibrillation with or without being guided by FIRMap (using RhythmView™ Workstation from TOPERA)
  Other Names: RFCA

SUMMARY:
Specific Aim: This prospective randomized study aims to compare the impact of three different catheter ablation approaches on long-term procedure outcome in terms of arrhythmia recurrence in persistent (PeAF) and long-standing persistent atrial fibrillation (LSPAF) patients. The three strategies to be evaluated are 1) ablation at sources guided by FIRMap (using RhythmView™ Workstation from TOPERA), 2) ablation at sources guided by FIRMap + conventional pulmonary vein antrum isolation (PVAI) and 3) Extended PVAI plus ablation of non-PV triggers and complex fractionated atrial electrograms (CFAE).

DETAILED DESCRIPTION:
Specific Aim: This prospective randomized study aims to compare the impact of three different catheter ablation approaches on long-term procedure outcome in terms of arrhythmia recurrence in persistent (PeAF) and long-standing persistent atrial fibrillation (LSPAF) patients. The three strategies to be evaluated are 1) ablation at sources guided by FIRMap (using RhythmView™ Workstation from TOPERA), 2) ablation at sources guided by FIRMap + conventional pulmonary vein antrum isolation (PVAI) and 3) Extended PVAI plus ablation of non-PV triggers and complex fractionated atrial electrograms (CFAE).

Hypothesis: Extended PVAI plus ablation of non-PV triggers and CFAE results in better long-term procedure outcome in PeAF and LSPAF patients.

Background: The limited success rate of conventional ablation approaches in LSPAF has led to the search for the ideal ablation strategy (1). The main problem in the settings of PeAF and LSPAF is the lack of information on the best targets to ablate to achieve freedom from arrhythmia (2). Some strategies aim at elimination of AF triggers; some solely target CFAE for atrial substrate modification whereas others elect for isolation of PVs plus posterior wall along with ablation of non-PV triggers demonstrated by high-dose isoproterenol challenge with or without CFAEs. (2). The last option has been shown to be the best option so far in improving the freedom from AF at long-term follow-up (2, 3).

Recently Narayan et al, by using a computational mapping system that identifies 'rotors' (organized reentrant circuits or focal impulses), were able to achieve a success rate of 82.4% following ablation of rotors plus PVAI, at a median follow-up of 273 days, in a primarily paroxysmal AF population (4). The results of this study are promising and need to be tested in patients with PeAF and LSPAF.

Objective: To compare the long-term efficacy and safety of different ablation approaches in PeAF and LSPAF patients.

Study Design: This prospective study will enroll 120 consecutive PeAF/LSPAF patients and consenting patients will be randomized to any of the 3 groups (40 per group); Group 1: ablation at sources guided by FIRMap (using RhythmView™ Workstation from TOPERA) Group 2: ablation at sources guided by FIRMap + conventional pulmonary vein antrum isolation (PVAI) Group 3: Extended PVAI plus ablation of non-PV triggers and complex fractionated atrial electrograms (CFAE) Patients will be randomized to different treatment groups after the risks and benefits of each one are discussed in detail with them.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years
2. Patients presenting with persistent or long-standing persistent AF
3. Undergoing first ablation procedure
4. Ability to provide written informed consent

Exclusion Criteria:

1. Reversible causes of atrial arrhythmia such as hyperthyroidism, pneumonia, pulmonary embolism, sarcoidosis and excessive alcohol consumption
2. Prior ablation procedures
3. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Recurrence of atrial arrhythmia | 1 year post-ablation
  Any episode of AF/AT > 30 sec will be considered as a recurrence. Episodes that occur during the first 2 months after the procedure (blanking period) will not be considered as recurrence.

SECONDARY OUTCOMES:
Procedural complications | 48 hours
  complications associated with prolonged use of radiofrequency (RF) energy such as atrioesophageal fistula, perforation, cardiac tamponade, major hemorrhagic events
Acute success | Intra-procedural
  AF termination, organization into AT or ≥10 % slowing

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Study Director — Texas Cardiac Arrhythmia Research Foundation
Locations (1):
- Texas Cardiac Arrhythmia Institute, St. david's Medical Center, Austin, Texas, United States

REFERENCES:
- [Derived] Mohanty S, Gianni C, Trivedi C, Metz T, Bai R, Al-Ahmad A, Bailey S, Burkhardt JD, Gallinghouse GJ, Horton R, Hranitzky PM, Sanchez JE, Di Biase L, Natale A. Impact of rotor ablation in non-paroxysmal AF patients: Findings from the per-protocol population of the OASIS trial at long-term follow-up. Am Heart J. 2018 Nov;205:145-148. doi: 10.1016/j.ahj.2018.05.021. Epub 2018 Jul 31. PMID 30144981
- [Derived] Mohanty S, Gianni C, Mohanty P, Halbfass P, Metz T, Trivedi C, Deneke T, Tomassoni G, Bai R, Al-Ahmad A, Bailey S, Burkhardt JD, Gallinghouse GJ, Horton R, Hranitzky PM, Sanchez JE, Di Biase L, Natale A. Impact of Rotor Ablation in Nonparoxysmal Atrial Fibrillation Patients: Results From the Randomized OASIS Trial. J Am Coll Cardiol. 2016 Jul 19;68(3):274-282. doi: 10.1016/j.jacc.2016.04.015. Epub 2016 May 6. PMID 27163758